CLINICAL TRIAL: NCT02070822
Title: Combination of Dynamic Contrast-enhanced and Diffusion-weighted Imaging and Magnetic Resonance Spectroscopy in 3T MRI to Early Predict Treatment Efficacy in Patients Receiving Transarterial Chemoembolization for Hepatocellular Carcinoma
Brief Title: 3T MRI to Predict TACE Response of HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201012077RB
Record Dates: First submitted 2012-01-02; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Magnetic resonance imaging
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TACE patients, for HCC: unresectable HCC patients

SUMMARY:
This study is a prospective clinical study using DCE-MRI, DWI and MRS in 3T scanner to evaluate tumors in patients with unresectable HCC after TACE. A total of 100 subjects will be recruited. MRI will be performed before TACE (day 0), day 14, and day 28 to assess the tumor responses. After day 28, all subjects will receive standard clinical care and be follow-up for 1 year. The imaging parameters will be compared among each MRI and correlate with patients' outcome. The investigators hypothesis that it might be helpful to combine DCE-MRI, DWI, and MRS for assessment of tumor response after TACE and predict patients' prognosis.

DETAILED DESCRIPTION:
Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) is a non-invasive quantitative technique for assessing micro-vascular structure by tracking the pharmacokinetics of injected low-molecular weight contrast agents as they pass through the tumor vasculature. This modality is being increasingly used in many oncological studies to characterize tumor angiogenesis and invasiveness, and monitor the treatment response.

Diffusion-weighted imaging (DWI) enables qualitative and quantitative assessment of tissue diffusivity (apparent diffusion coefficient, ADC) without the use of gadolinium chelates. DWI has been suggested to be useful in monitoring the response of HCC after TACE because of earlier assessment of tumor necrosis with increasing ADC values.

MR spectroscopy facilitates the study of cellular metabolism and in vivo detection of abnormalities. A few studies of in vivo MR spectroscopy reported an increase in choline levels within tumors such as HCC and a reduction in the lipid-to-choline ratio after conventional TACE was performed for HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Prior Informed Consent Form
2. Patients who had undergone surgery for the treatment of HCC are allowed.
3. At least one measurable tumor, according to RECIST version 1.1.
4. Age more than 20 years.
5. ECOG performance status 0 or 1.
6. Life expectancy more than 3 months.
7. Child-Pugh class A.
8. Unresectable, multinodular tumors
9. Confirmed Diagnosis of HCC
10. At least one uni-dimensional lesion measurable according to the Modified RECIST criteria by MRI
11. Adequate bone marrow, liver and renal function

Exclusion Criteria:

1. History of TACE
2. Diffuse infiltrative HCC or presence of main portal vein invasion or extrahepatic metastasis
3. Any contraindications for hepatic embolization procedures:, including hepatofugal blood flow, large intrahepatic or porto-systemic shunt, impaired clotting test, renal failure requiring hemo-or peritoneal dialysis
4. Any contraindication for MRI, including known contrast allergy, electronically operated implants or devices, and claustrophobia.
5. Other acute or chronic medical, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation and is inappropriate for this study by the judgment of the investigator
6. Known history of HIV infection
7. Concurrent primary extrahepatic cancer
8. Pregnant or breast-feeding subjects

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients, admitted for TACE treatment of HCC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
tumor response | change of tumor size from baseline to at 6 months
  change of tumor size from baseline to at 6 months

SECONDARY OUTCOMES:
change of baseline MRI parameters | change of MRI parameters from baseline to at 6 months
  comparsion of MRI parameters from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bang-Bin Chen, MD, Principal Investigator — National Taiwan Uinversity Hospital
Locations (1):
- National Taiwan Uinversity Hospital, Taipei, Taipei, Taiwan